CLINICAL TRIAL: NCT02524028
Title: Relationship Between Autonomic Central Nervous System Activation and Atrial Fibrillation: A Prospective Functional MRI Study (fMRI)
Brief Title: Relationship Between Autonomic Central Nervous System Activation and Atrial Fibrillation Using Functional MRI (fMRI)
Acronym: fMRI
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Nassir F. Marrouche, MD, Associate Professor, University of Utah
Other Study IDs: IRB_00044089
Record Dates: First submitted 2013-09-17; First posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; fMRI
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case Participant Cohort: Participants with atrial fibrillation
- Control Participant Cohort: Participants without atrial fibrillation or any other heart disease

SUMMARY:
The fMRI study is a prospective study with the objective of evaluating the effects of the autonomic central nervous system on the regulation of heart rate in patients with atrial fibrillation (AF). This study will compare a functional MRI (fMRI) scan in patients prior to a direct current cardioversion (DCCV) to a second fMRI scan taken post DCCV. In addition, this study will compare functional MRI (fMRIs) to a control group of heart healthy, age-matched patients who will also receive two fMRI scans spaced about one week apart.

Our expectation is that at the end of this study, the investigators will have greater insight into the role of the central nervous system and more specifically the autonomic nervous system in modulating AF. The investigators expect that understanding the interaction between the central nervous system and cardiac arrhythmias will lead to the development of novel therapies that preserve and restore normal sinus rhythm. This study will serve as a pilot study with the goal of obtaining additional grant funding and expanding the study once differences in volumes of activation are demonstrated.

DETAILED DESCRIPTION:
The central nervous system (CNS) consists of the brain and spinal cord and serves as the collection point of nerve impulses. The peripheral nervous system (PNS) includes all nerves not in the brain or spinal cord and connects all parts of the body to the CNS. The autonomic nervous system (ANS), which consists mostly motor nerves, controls functions of involuntary smooth muscles, glands, and cardiac muscles. The ANS is further divided into the sympathetic and parasympathetic systems. In relation to the heart, the sympathetic system controls increases in heart rate, blood pressure, and cardiac output. The parasympathetic system lowers heart activity and operates during normal situations where the body is not under stress1, 2.

While the influence of the central nervous system on cardiac rhythm and function is well accepted, the mechanisms of this control are poorly understood. A preponderance of data implicates the autonomic nervous system in the development of many cases of atrial fibrillation (AF)3, 4. The importance of investigating the role of the central nervous system in the control of the heart rhythm can be appreciated when reviewing the prevalence of cardiac arrhythmias. AF alone affects 2.2 million adults in the United States. With the growing aged population, this number can be expected to rise to 5.6-10 million by the year 2050. AF contributes to the development of heart failure and stroke and can precipitate angina in some patients. New therapies are needed since both surgical and minimally invasive ablative techniques are associated with a substantial failure rate in addition to the complications of invasive procedures. Understanding the CNS's role promises to direct new therapies to improve treatment success and reduce complications associated with therapy for AF and other arrhythmias.

Direct current (DC) cardioversion (DCCV) is a procedure in which a synchronized electrical shock is delivered through the chest to the heart via electrodes that are applied to the skin of the chest and back. Most elective cardioversion procedures are performed to treat AF or atrial flutter (AFL). The shock causes all the heart cells to contract simultaneously, thereby interrupting and terminating the abnormal electrical rhythm of AF without damaging the heart. This interruption of the abnormal beat allows the electrical system in the heart to regain control and restore a normal sinus rhythm (see Figure 1, Appendix A). Since the shock can be painful, the patient is usually sedated. Once sedated, the physician charges the defibrillator to a specified energy level and then delivers the shock. Additional shocks at higher energy levels can be delivered if the first attempt does not restore sinus rhythm. Typically patients are able to go home about an hour after the procedure. DCCV will restore normal sinus rhythm in 90% of patients5.

Newer MRI techniques offer the ability to not only image anatomy, but also to assess brain activation patterns. Functional magnetic resonance imaging (fMRI) was developed in the early 1990s, and is a variation of magnetic resonance imaging (MRI). The primary purpose of fMRI is to observe brain function under varying stimuli in a non-invasive way. fMRI uses a conventional MRI scanner. It takes advantage of the magnetic properties of iron in the blood. Whenever any part of the brain becomes active, the small blood vessels in that localized region dilate, causing more blood to rush into that region of the brain. The blood's iron atoms cause small distortions in the magnetic field around them, which causes the MRI scanner to be able to read and display an image of the brain's activity. When a region of the brain is activated, a large amount of freshly oxygenated blood pours into that structure of the brain, thus causing a small change in the magnetic field, and producing an MRI signal in the active region6.

Prior studies have utilized heart rate variation or galvanic skin response as an independent measure of autonomic arousal and compared these measures to fMRI to determine regions of the brain that are active during sympathetic or parasympathetic arousal 7-11. Studies have typically identified activation within the anterior cingulate region and insular cortex during sympathetic activation and in the ventral anterior cingulate in parasympathetic activation12, 13. Moreover, attenuation of the parasympathetic myocardial innervations by myocardial fat pad or ablation of parasympathetic ganglionic plexi have been shown to suppress AF in a significant number of patients presenting with this arrhythmia14, 15. Whether attenuation of the central autonomic pathways plays a role in initiating AF, or if atrial arrhythmias may lead to this central attenuation is an open question. This study is aimed at defining the effect of AF on the central autonomic pathways and vise versa.

Our expectation is that at the end of this study, we will have greater insight into the role of the central nervous system and more specifically the autonomic nervous system in modulating AF. We expect that understanding the interaction between the central nervous system and cardiac arrhythmias will lead to the development of novel therapies that preserve and restore normal sinus rhythm.

This study will serve as a pilot study with the goal of obtaining additional grant funding and expanding the study once differences in volumes of activation are demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* AF patients presenting for DCCV
* Right-handed

Exclusion Criteria:

* Any neuropsychiatric illness, including substance abuse.
* Any medical or neurological disease likely to impact the central nervous system.
* Subject has a metal implant, pacemaker or other contraindication for MRI or fMRI.
* Currently being treated with any medication that affects the central nervous system.
* Women currently pregnant, breastfeeding or of childbearing age not currently taking or not willing to use a reliable form of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential participants for the fMRI Study will be recruited from the Cardiology/Electrophysiology (EP) clinic during normally scheduled clinic visits. Control participants will be recruited from other hospital clinics.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pre- and post- cardioversion fMRI scans will be compared | fMRI pre cardioversion and fMRI within a week of cardioversion

CONTACTS AND LOCATIONS:
Overall Officials: Nassir F Marrouche, MD, FHRS, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States